CLINICAL TRIAL: NCT03016754
Title: Heart Failure Optimization Study
Acronym: HF-Opt
Status: Completed | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90D0109
Record Dates: First submitted 2017-01-04; First posted 2017-01-11 (Estimated); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Sudden Cardiac Death; Sudden Cardiac Arrest; Heart Failure; Heart Failure Low Output
Keywords: sudden cardiac death (SCD); sudden cardiac arrest (SCA); heart failure (HF); heart failure with reduced ejection fraction (HFrEF); guideline directed medical therapy (GDMT); guideline recommended medical therapy (GRMT); wearable cardioverter defibrillator (WCD)
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Early Recovery: Patients improved to LVEF >35% within the first 90 days following GDMT. These patients are expected to end WCD use and not receive an implantable cardioverter defibrillator (ICD) according to current guidelines.
- Improvement: Patients improved LVEF from start of WCD use (a positive change of at least 5% in LVEF) or have borderline LVEF of 30-35% at day 90. These patients were expected, but not required to continue to use the WCD for an additional 90 days.
  Interventions: Device: Wearable Cardioverter Defibrillator
- Non-improvement: Patients show no change, worsening of LVEF or LVEF <30%. Those on GDMT are expected to be evaluated for an ICD. Those not yet on GDMT were expected, but not required, to continue the WCD for an additional 90 days.
  Interventions: Device: Wearable Cardioverter Defibrillator

INTERVENTIONS:
Device: Wearable Cardioverter Defibrillator — LifeVest is the brand of Wearable Cardioverter Defibrillator used in this study.
  Other Names: LifeVest
  Groups: Improvement; Non-improvement

SUMMARY:
This study is designed as a multi-center prospective observational study of newly diagnosed Heart Failure (HF) patients to test the hypothesis that additional Ejection Fraction (EF) recovery occurs between 90 and 180 days as Guideline Directed Medical Therapy (GDMT) is achieved. Although the study doesn't start until day 90, all eligible, consenting patients will be entered into a registry at the start of wearable cardioverter defibrillator (WCD) use. The pre-study registry will allow us to collect early (90 day) outcomes and data in those patients who are likely to be eligible for the study at day 90, or are eligible, but refuse the study at day 90.

DETAILED DESCRIPTION:
This study will be conducted at thirty to sixty sites, initially in US and Europe. It will be used to observe the rate of recovery of ventricular function (EF>35%) between 90 and 180 days in newly diagnosed HF patients who were prescribed the WCD ≤ 10 days post-discharge after hospitalization for a primary reason of new onset HF (≤30 days since first HF hospitalization), with ischemic or non-ischemic cardiomyopathy, and have already used a WCD for 90 ± 14 days. For the first 90 days of WCD use, patients will be enrolled in a pre-study registry. The FDA-approved WCD will be prescribed for up to 6 months of use after hospital discharge, with the option for longer use under physician discretion. Approximately 870 subjects will enroll into the pre-study registry and 750 subjects into the study.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 (Registry phase)

* Patients (≥18 years old) who were prescribed the WCD ≤ 10 days post-discharge after hospitalization for a primary reason of new onset HF (≤30 days since first HF hospitalization), with ischemic or nonischemic cardiomyopathy, and have used the WCD for no more than 30 days.
* Patients who had an EF ≤ 35% during index hospitalization (must be last measurement if performed multiple times).

Phase 2 (Study phase)

* Patients who completed Phase 1 and used a WCD for 90 ± 14 days.

Exclusion Criteria (both phases):

* Patients under 18 years old.
* Patients who have an active unipolar pacemaker.
* Patients with a physical or mental condition that could impair their ability to properly interact with the device.
* Patients currently participating in another clinical study.
* Patients with any skin condition that would prevent wearing the device.
* Patients with an advanced directive prohibiting resuscitation.

Exclusion criteria (Phase 2)

* Patients who have a QRS duration of ≥135 ms and are planned for cardiac resynchronization therapy.
* Patients with recent myocardial infarction or coronary revascularization (since start of WCD wear; i.e. 0-90 days of WCD wear).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (≥18 years old) who used a WCD for 90 days after hospitalization for a primary reason of new onset HF with ischemic or nonischemic cardiomyopathy.
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Osz, Study Director — Director, Clinical Operations
Locations (67):
- United States (39):
  - UAB Division of Cardiovascular Disease, Birmingham, Alabama
  - Study Site, West Hills, California
  - Baptist Heart Specialists, Fernandina Beach, Florida
  - Baptist Heart Specialists, Jacksonville, Florida
  - Baptist Heart Specialists, Jacksonville Beach, Florida
  - Institute of Cardiovascular Research, Ocala, Florida
  - Research Physicians Network Alliance, Orlando, Florida
  - Study Site, St. Petersburg, Florida
  - Fox Valley Clinical Research Center, Aurora, Illinois
  - Chicago Medical Research, LLC, Hazel Crest, Illinois
  - Unity Point Health-Methodist, Peoria, Illinois
  - Cardiovascular Research of Northwest Indiana, LLC, Munster, Indiana
  - Beacon Medical Group clinical Research, South Bend, Indiana
  - Saint Joseph London, London, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Covenant Medical Center, Inc., Saginaw, Michigan
  - Jackson Heart Clinic, Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - SSM Health Heart & Vascular, Lake Saint Louis, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Hackensack Meridian Health, Hackensack, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Trinity Medical Center, Buffalo, New York
  - SJH Cardiology, Liverpool, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - City Cardiology Associates, Barberton, Ohio
  - Drexel University, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Guthrie Medical Group, P.C., Sayre, Pennsylvania
  - Carolina Heart Specialists, Lancaster, South Carolina
  - Sanford Health, Sioux Falls, South Dakota
  - Methodist University Hospital (MUH) and Methodist OliveBranch (MOB), Memphis, Tennessee
  - Methodist South (MS) University Hospital, Memphis, Tennessee
  - Parkway Cardiology, Oak Ridge, Tennessee
  - Texas Health Research & Education Institute, Dallas, Texas
  - Mission Research Insitute, New Braunfels, Texas
  - Providence Health Center, Waco, Texas
  - St. Mary's Medical Center, Huntington, West Virginia
- Austria (2):
  - Ordensklinikum Linz GmbH/Elisabethinen, Linz
  - Medizinische Universitätsklinik Wien, Vienna
- France (6):
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHU de Grenoble site Nord- Hopital Albert Michallon, Grenoble
  - CHU de Clermont-Ferrand- Hopital Albert Michallon, Grenoble
  - Hopital Europeen Georges Pompidou, Paris
  - CHU Pontchaillou, Rennes
  - Clinique Pasteur, Toulouse
- Germany (20):
  - Amper Kliniken AG, Heliios Amper-Klinikum Dachau, Dachau, Bavaria
  - Klinik u. Polikllinik Fur Innere Med. II Kardiologie, Regensburg, Bavaria
  - Schwarzwald-Baar Klinik, Villingen-Schwenningen, Deutschland
  - Elisabeth-Krankenhaus, Essen, North Rhine-Westphalia
  - Klinikum Augsburg, Augsburg
  - Herz- und Gefäßklinik Bad Neustadt, Bad Neustadt an der Saale
  - Asklepios Klinik Barmbek, Barmbek
  - Charité Universitätsmedizin Berlin, Berlin
  - St. Vinzenz Hospital, Cologne
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - UKGM, Standort Giessen, Giessen
  - Asklepios Harzklinik Goslar, Goslar
  - Universitatsklinikum Halle, Halle
  - Asklepios Klinik Wandsbek, Hamburg
  - Kardiologie, Asklepios Klinik St. Georg, Hamburg
  - Medizinische Hochschule Hannover, Hannover
  - Herzzentrum Leipzig GmbH, Leipzig
  - Klinikum Ludenscheid, Lüdenscheid
  - Katholisches Klinikum Lunen, Lünen
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were initially screened from the prescribed wearable cardioverter defibrillator (WCD) patients and enrolled into a pre-study registry (n=1300). At 90 +/- 14 days of WCD use, patients were screened from the site's pre-study registry participants. Subjects determined to be ineligible for the study or those exiting the registry before study phase were excluded (n=698). The study phase started at day 90.
Groups:
- Early Recovery: Patients improved to LVEF >35% within the first 90 days following guideline directed medical therapy (GDMT). These patients are expected to end wearable cardioverter defibrillator (WCD) use and not receive an implantable cardioverter defibrillator (ICD) according to current guidelines.
- Improvement: Patients improved LVEF from start of WCD use (a positive change of at least 5% in LVEF) or have borderline LVEF of 30-35% at day 90. These patients were expected, but not required to continue to use the WCD for an additional 90 days.
  Wearable Cardioverter Defibrillator: LifeVest Wearable Cardioverter Defibrillator
- Non-improvement: Patients show no change, worsening of LVEF or LVEF <30%. Those on guideline directed medical therapy (GDMT) are expected to be evaluated for an implantable cardioverter defibrillator (ICD). Those not yet on GDMT were expected, but not required, to continue the WCD for an additional 90 days.
  Wearable Cardioverter Defibrillator: LifeVest Wearable Cardioverter Defibrillator
- Unassigned Based on Left Ventricular Ejection Fraction (LVEF): Study subjects missing a day 90 LVEF value and were unable to be assigned to a group.
Period: Overall Study
Arm/Group | Early Recovery | Improvement | Non-improvement | Unassigned Based on Left Ventricular Ejection Fraction (LVEF)
Started | 279 | 214 | 90 | 19
Completed | 243 | 183 | 77 | 9
Not Completed | 36 | 31 | 13 | 10
Not completed — Death | 5 | 4 | 5 | 1
Not completed — Lost to Follow-up | 23 | 17 | 4 | 2
Not completed — Withdrawal by Subject | 6 | 6 | 2 | 2
Not completed — Other/Unknown | 2 | 4 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Subjects consented and enrolled into the study phase at Day 90.
Groups:
- Early Recovery: Patients improved to LVEF >35% within the first 90 days following guideline directed medical therapy (GDMT). These patients are expected to end WCD use and not receive an implantable cardioverter defibrillator according to current guidelines.
- Non-improvement: Patients show no change, worsening of LVEF or LVEF <30%. Those on guideline directed medical therapy (GDMT) are expected to be evaluated for an implantable cardioverter defibrillator. Those not yet on GDMT were expected, but not required, to continue the WCD for an additional 90 days.
- Total: Total of all reporting groups
Arm/Group | Early Recovery | Improvement | Non-improvement | Unassigned Based on Left Ventricular Ejection Fraction (LVEF) | Total
Number analyzed (Participants) | 279 | 214 | 90 | 19 | 602
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13) | 57 (14) | 60 (13) | 58 (11) | 59 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 49 | 25 | 2 | 164
  Male | 191 | 165 | 65 | 17 | 438
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian or Alaskan native | 2 | 1 | 0 | 1 | 4
  Race/Ethnicity: Asian | 0 | 2 | 1 | 0 | 3
  Race/Ethnicity: Caucasian | 231 | 173 | 65 | 15 | 484
  Race/Ethnicity: Hispanic or Latin | 4 | 3 | 5 | 0 | 12
  Race/Ethnicity: Black or African American | 31 | 27 | 15 | 2 | 75
  Race/Ethnicity: Other | 0 | 0 | 1 | 0 | 1
  Race/Ethnicity: No response | 7 | 8 | 3 | 1 | 19
  Race/Ethnicity: Multiple races selected | 4 | 0 | 0 | 0 | 4
Region of Enrollment [Number; unit: participants]
  Austria | 10 | 1 | 1 | 4 | 16
  United States | 151 | 115 | 57 | 8 | 331
  France | 3 | 6 | 2 | 4 | 15
  Germany | 115 | 92 | 30 | 3 | 240
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.0 (7.4) | 29.0 (6.4) | 29.8 (7.2) | 28.7 (6.2) | 29.6 (7.0)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 124 (22) | 116 (19) | 118 (15) | 124 (20) | 120 (20)
History of hypertension (HTN) [Count of Participants; unit: Participants] | 196 | 122 | 54 | 14 | 386
History of diabetes [Count of Participants; unit: Participants] | 69 | 61 | 27 | 7 | 164
History of chronic obstructive pulmonary disease (COPD) [Count of Participants; unit: Participants] | 37 | 17 | 17 | 0 | 71
History of transient ischemic attack/Cerebrovascular accident [Count of Participants; unit: Participants] | 18 | 18 | 5 | 1 | 42
History of chronic kidney disease [Count of Participants; unit: Participants] | 29 | 24 | 11 | 2 | 66
Ischemic cardiomyopathy [Count of Participants; unit: Participants] | 113 | 70 | 39 | 8 | 230
Non-ischemic cardiomyopathy [Count of Participants; unit: Participants] | 156 | 135 | 47 | 10 | 348
Mixed cardiomyopathy [Count of Participants; unit: Participants] | 10 | 9 | 4 | 1 | 24
History of sudden cardiac arrest [Count of Participants; unit: Participants] | 7 | 3 | 7 | 1 | 18
History of arrhythmia in past year [Count of Participants; unit: Participants]
  Atrial Flutter | 14 | 8 | 0 | 2 | 24
  Atrial fibrillation | 68 | 31 | 12 | 2 | 113
  Sinus tachycardia | 35 | 36 | 14 | 0 | 85
  Supraventricular tachycardia | 6 | 5 | 2 | 0 | 13
  Ventricular tachycardia | 8 | 2 | 1 | 2 | 13
  Ventricular fibrillation | 1 | 0 | 0 | 0 | 1
  Ventricular tachycardia (non-sustained | 9 | 11 | 8 | 1 | 29
  Sinus bradycardia | 5 | 3 | 2 | 0 | 10
  First-degree AV block | 2 | 4 | 0 | 1 | 7
  Type I Second-degree AV block | 0 | 1 | 0 | 0 | 1
  Type II Second-degree AV block | 0 | 1 | 0 | 0 | 1
  Third degree AV block | 0 | 1 | 0 | 0 | 1
  Paced rhythm | 0 | 3 | 0 | 0 | 3
Initial heart rate [Mean (Standard Deviation); unit: Beats per minute] | 80 (17) | 84 (18) | 85 (16) | 74 (23) | 82 (18)
Initial respiration rate [Mean (Standard Deviation); unit: Breaths per minute] | 17 (3) | 17 (3) | 17 (3) | 16 (2) | 17 (3)
History of myocardial infarction [Count of Participants; unit: Participants] | 66 | 30 | 28 | 5 | 129
History of coronary artery bypass graft surgery [Count of Participants; unit: Participants] | 25 | 15 | 9 | 3 | 52
History of percutaneous coronary intervention [Count of Participants; unit: Participants] | 71 | 34 | 23 | 6 | 134
New York Heart Association (NYHA) functional class at index hospitalization [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification places patients in 1 of 4 categories based on limitations of physical activity. The healthcare practitioner assigns the patient at baseline and then again at follow-ups.
  I= No limitation of physical activity. II= Slight limitation of physical activity. III= Marked limitation of physical activity. IV= Symptoms of heart failure at rest- Any physical activity causes further discomfort.
  Participants
    Class I | 7 | 6 | 0 | 1 | 14
    Class II | 56 | 40 | 16 | 3 | 115
    Class III | 100 | 77 | 41 | 6 | 224
    Class IV | 31 | 26 | 7 | 2 | 66
    Not documented | 85 | 65 | 26 | 7 | 183
New York Heart Association (NYHA) functional class at registry start [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification places patients in 1 of 4 categories based on limitations of physical activity. The healthcare practitioner assigns the patient at baseline and then again at follow-ups.
  I= No limitation of physical activity. II= Slight limitation of physical activity. III= Marked limitation of physical activity. IV= Symptoms of heart failure at rest- Any physical activity causes further discomfort.
  Participants
    Class I | 17 | 11 | 3 | 3 | 34
    Class II | 85 | 70 | 26 | 3 | 184
    Class III | 68 | 37 | 27 | 5 | 137
    Class IV | 5 | 3 | 1 | 0 | 9
    Not documented | 104 | 93 | 33 | 8 | 238

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With LVEF Recovery at Day 90 and 180
Description: The percentage of patients reaching the goal of LVEF>35% will be compared at 90 days and 180 days. Echocardiographic assessment of LVEF was used.
Time Frame: 180 days
Population: Subjects with all three LVEF measurements (baseline, day 90, day 180) were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Non-improvement: Patients show no change, worsening of LVEF or LVEF <30%. Those on guideline directed medical therapy (GDMT) are expected to be evaluated for an implantable cardioverter defibrillator. Those not yet on GDMT were expected, but not required, to continue the WCD for an additional 90 days.
  Wearable Cardioverter Defibrillator: LifeVest Wearable Cardioverter Defibrillator
Arm/Group | Early Recovery | Improvement | Non-improvement
Number analyzed (Participants) | 222 | 186 | 79
Participants
  Day 90 LVEF: Day 90 LVEF >35% | 222 | 0 | 0
  Day 90 LVEF: Day 90 LVEF <=35% | 0 | 186 | 79
  Day 180 LVEF: Day 90 LVEF >35% | 208 | 97 | 25
  Day 180 LVEF: Day 90 LVEF <=35% | 14 | 89 | 54

2. Primary Outcome: Percentage of Study Subjects Reaching Target Doses of Guideline Directed Medical Therapy (GDMT)
Description: Descriptive statistics will be used to assess the percentage of study subjects reaching target doses of GDMT at 90 and 180 days. All eligible study subjects with LVEF data at all three timepoints were used for this analysis.
Time Frame: 180 days
Population: Subjects with all three LVEF measurements (baseline, day 90, day 180) were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Recovery | Improvement | Non-improvement
Number analyzed (Participants) | 222 | 186 | 79
Participants
  Reached target dose beta-blocker at Day 90: Target dose reached | 57 | 36 | 16
  Reached target dose beta-blocker at Day 90: Target dose not reached | 164 | 149 | 63
  Reached target dose beta-blocker at Day 90: Dose not available | 1 | 1 | 0
  Reached target dose RAS antagonist at Day 90: Target dose reached | 86 | 59 | 16
  Reached target dose RAS antagonist at Day 90: Target dose not reached | 136 | 125 | 63
  Reached target dose RAS antagonist at Day 90: Dose not available | 0 | 2 | 0
  Reached target dose mineralocorticoid receptor antagonist at Day 90: Target dose reached | 114 | 77 | 30
  Reached target dose mineralocorticoid receptor antagonist at Day 90: Target dose not reached | 108 | 109 | 49
  Reached target dose mineralocorticoid receptor antagonist at Day 90: Dose not available | 0 | 0 | 0
  Reached target dose beta-blocker at Day 180: Target dose reached | 56 | 47 | 19
  Reached target dose beta-blocker at Day 180: Target dose not reached | 166 | 139 | 60
  Reached target dose beta-blocker at Day 180: Dose not available | 0 | 0 | 0
  Reached target dose RAS antagonist at Day 180: Target dose reached | 92 | 84 | 22
  Reached target dose RAS antagonist at Day 180: Target dose not reached | 130 | 101 | 56
  Reached target dose RAS antagonist at Day 180: Dose not available | 0 | 1 | 1
  Reached target dose mineralocorticoid receptor antagonist at Day 180: Target dose reached | 103 | 84 | 30
  Reached target dose mineralocorticoid receptor antagonist at Day 180: Target dose not reached | 119 | 102 | 49
  Reached target dose mineralocorticoid receptor antagonist at Day 180: Dose not available | 0 | 0 | 0

3. Secondary Outcome: All Subjects With Sustained Ventricular Tachycardia (VT)/Ventricular Fibrillation (VF) Arrhythmias During WCD Use
Description: Observe the percentage of patients having sustained VT/VF arrhythmias during WCD use. As this was a secondary outcome to describe events during all WCD use, all eligible registry subjects were used for this analysis. Participants were not split into groups for secondary analyses, only for reporting results of left ventricular ejection fraction (LVEF) recovery in the primary outcomes.
Time Frame: 360 days
Population: Subjects consented and enrolled into the study phase at Day 90.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Recovery | Improvement | Non-improvement | Unassigned Based on Left Ventricular Ejection Fraction (LVEF)
Number analyzed (Participants) | 279 | 214 | 90 | 19
Participants | 4 | 1 | 0 | 0

4. Secondary Outcome: All Sustained Ventricular Tachycardia (VT)/Ventricular Fibrillation (VF) Arrhythmias Events During WCD Use
Description: Observe the occurrence of all sustained VT/VF arrhythmias during WCD use by event. As this was a secondary outcome to describe events during all WCD use, all eligible registry subjects were used for this analysis. Participants were not split into groups for secondary analyses, only for reporting results of left ventricular ejection fraction (LVEF) recovery in the primary outcomes.
Time Frame: 360 days
Population: Subjects consented and enrolled into the study phase at Day 90.
Measure: Number; unit: events
Arm/Group | Early Recovery | Improvement | Non-improvement | Unassigned Based on Left Ventricular Ejection Fraction (LVEF)
Number analyzed (Participants) | 279 | 214 | 90 | 19
events | 5 | 1 | 0 | 0

5. Secondary Outcome: Percentage of All Patients Having Other Arrhythmias
Description: Observe the percentage of patients having other arrhythmias during WCD use, such as asystole and supra-ventricular arrhythmias that are recorded by the device. As this was a secondary outcome to describe events during all WCD use, all eligible registry subjects were used for this analysis. Participants were not split into groups for secondary analyses, only for reporting results of left ventricular ejection fraction (LVEF) recovery in the primary outcomes.
Time Frame: 180 days
Population: Subjects consented and enrolled into the study phase at Day 90.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Recovery | Improvement | Non-improvement | Unassigned Based on Left Ventricular Ejection Fraction (LVEF)
Number analyzed (Participants) | 279 | 214 | 90 | 19
Participants
  Asystole | 0 | 1 | 0 | 0
  Non-sustained ventricular tachycardia | 0 | 1 | 2 | 0
  Supraventricular tachycardia | 13 | 20 | 4 | 1
  Sinus tachycardia | 1 | 0 | 0 | 0

6. Secondary Outcome: Efficacy in Treating Ventricular Arrhythmias
Description: Observe the effectiveness of the wearable cardioverter defibrillator worn by this population in treating ventricular arrhythmias. As this was a secondary outcome to describe events during all WCD use, all eligible registry subjects were used for this analysis. Participants were not split into groups for secondary analyses, only for reporting results of left ventricular ejection fraction (LVEF) recovery in the primary outcomes.
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Groups:
- All Registry Subjects With Appropriate Shock for VT/VF: Clinical outcomes and device data from any defibrillation or cardiac event will be reviewed for success as defined by appropriate detection and defibrillation, conversion out of the detected ventricular arrhythmia, and consciousness when medically evaluated after treatment.
Arm/Group | All Registry Subjects With Appropriate Shock for VT/VF
Number analyzed (Participants) | 7
Participants
  Successfully cardioverted by the wearable cardioverter defibrillator | 7
  Not successfully cardioverted by the wearable cardioverter defibrillator | 0

7. Secondary Outcome: Mortality Analysis
Description: Evaluate the effect of wearable defibrillators on 180, 270, and 360-day mortality following discharge in HF patients. Cumulative assessment of survival will be made at these time points for those entered into the study (e.g. up to 180, 270, 360 days, or >360 days (up to 14 months)). A mortality review will be conducted by independent adjudicators to group all deaths as cardiac or non-cardiac, and sudden or non-sudden. All eligible study subjects were used for this analysis. Participants were not split into groups for secondary analyses, only for reporting results of left ventricular ejection fraction (LVEF) recovery in the primary outcomes. Data collected on deaths after the prespecified final timepoint (n=3) will be labeled >360 days (up to 14 months). 1 subject completed the study immediately prior to the reported death, hence the different number from the participant flow.
Time Frame: 0 to180, 0 to 270, and 0 to 360 days, or >360 days (up to 14 months)
Population: All patients in the Study were assessed for survival at Day 180, 270, and 360, or >360 days (up to 14 months). Patients who died were adjudicated for cause of death.
Measure: Count of Participants; unit: Participants
Groups:
- All Study Phase Subjects Who Died: All eligible Study phase subjects enrolled at Day 90 who died during follow-up
Arm/Group | All Study Phase Subjects Who Died
Number analyzed (Participants) | 16
Participants
  180 Day cumulative mortality: number analyzed (Participants) | 5
  180 Day cumulative mortality: Cardiovascular death_Sudden | 2
  180 Day cumulative mortality: Cardiovascular death_Non sudden | 1
  180 Day cumulative mortality: Non-cardiovascular death_Sudden | 1
  180 Day cumulative mortality: Non-cardiovascular death_Non Sudden | 0
  180 Day cumulative mortality: Unknown death_Sudden | 1
  180 Day cumulative mortality: Unknown death_Non Sudden | 0
  270 Day cumulative mortality: number analyzed (Participants) | 9
  270 Day cumulative mortality: Cardiovascular death_Sudden | 2
  270 Day cumulative mortality: Cardiovascular death_Non sudden | 2
  270 Day cumulative mortality: Non-cardiovascular death_Sudden | 1
  270 Day cumulative mortality: Non-cardiovascular death_Non Sudden | 3
  270 Day cumulative mortality: Unknown death_Sudden | 1
  270 Day cumulative mortality: Unknown death_Non Sudden | 0
  360 Day cumulative mortality: number analyzed (Participants) | 13
  360 Day cumulative mortality: Cardiovascular death_Sudden | 3
  360 Day cumulative mortality: Cardiovascular death_Non sudden | 2
  360 Day cumulative mortality: Non-cardiovascular death_Sudden | 1
  360 Day cumulative mortality: Non-cardiovascular death_Non Sudden | 6
  360 Day cumulative mortality: Unknown death_Sudden | 1
  360 Day cumulative mortality: Unknown death_Non Sudden | 0
  >360 Day cumulative mortality (up to 14 months): Cardiovascular death_Sudden | 3
  >360 Day cumulative mortality (up to 14 months): Cardiovascular death_Non sudden | 2
  >360 Day cumulative mortality (up to 14 months): Non-cardiovascular death_Sudden | 1
  >360 Day cumulative mortality (up to 14 months): Non-cardiovascular death_Non Sudden | 9
  >360 Day cumulative mortality (up to 14 months): Unknown death_Sudden | 1
  >360 Day cumulative mortality (up to 14 months): Unknown death_Non Sudden | 0

8. Secondary Outcome: Healthcare utilization_type
Description: Healthcare utilization (emergency room visits, hospitalizations, doctor visits etc.) on all patients during the period of the study. All eligible study subjects were used for this analysis. Participants were not split into groups for secondary analyses, only for reporting results of left ventricular ejection fraction (LVEF) recovery in the primary outcomes.
Time Frame: 360 days
Population: Healthcare utilization events (emergency room visits, hospitalizations, doctor visits etc.) for all patients during the period of the study.
Measure: Count of Units; unit: Heathcare Utilization Events
Units Other Than Participants: Heathcare Utilization Events
Groups:
- All Eligible Study Subjects: 598 study phase subjects were eligible for analysis.
Arm/Group | All Eligible Study Subjects
Number analyzed (Participants) | 598
Number analyzed (Heathcare Utilization Events) | 3130
Heathcare Utilization Events
  Doctor visits | 2640
  Hospitalizations | 247
  Emergency room visits | 125
  UrgiCare visits | 21
  Skilled nursing facility/rehabilitation | 16
  Observational stay | 81

9. Secondary Outcome: Healthcare utilization_length of Use
Description: Length of stay for any hospitalization, observation, skilled nursing facility stays. All eligible study subjects reporting one of these stays were used for this analysis, and grouped by type of stay. Participants were not split into groups for secondary analyses, only for reporting results of left ventricular ejection fraction (LVEF) recovery in the primary outcomes.
Time Frame: 360 days
Population: Events included Hospital, Observation, and skilled nursing facility stays
Measure: Median (Full Range); unit: days
Units Other Than Participants: Heathcare Utilization Events
Groups:
- Hospital Stays: Under the types of healthcare encounters, all the Hospital stays were analyzed for length of use.
- Observation Stays: Under the types of healthcare encounters, all the Observation stays were analyzed for length of use.
- Skilled Nursing Facility Stays: Under the types of healthcare encounters, all the Skilled nursing facility stays were analyzed for length of use.
Arm/Group | Hospital Stays | Observation Stays | Skilled Nursing Facility Stays
Number analyzed (Participants) | 171 | 61 | 9
Number analyzed (Heathcare Utilization Events) | 247 | 81 | 16
days | 3 [0 to 49] | 1 [0 to 15] | 2 [1 to 22]

10. Other Pre Specified Outcome: Complications From Extended Use
Description: The safety objectives will be to compare complications from extended use of the WCD with those of the ICD during the study phase timeframe. All eligible study subjects were used for this safety analysis. Participants were not split into groups for secondary analyses, only for reporting results of left ventricular ejection fraction (LVEF) recovery in the primary outcomes.
Time Frame: 360 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Eligible Study Subjects
Number analyzed (Participants) | 598
Participants
  Inappropriate shock from WCD during study phase (extended use >104 days) | 1
  Inappropriate shock from ICD during study phase | 0
  No reported inappropriate shock during study phase | 597

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed up to 14 months; serious and other (not including serious) adverse events were assessed for up to 1 year.
Description: All deaths, Serious Adverse Events, and Other Adverse Events are reported below. All adverse device effects (ADE) were classified by the investigator as anticipated or unanticipated. An unanticipated ADE is any adverse effect not identified by nature, severity, or frequency prior to the study.
  Commonly reported ADEs in patients having HF were not reported unless deemed to be related to WCD wear.
  Inappropriate shocks exceeding 3 per 100 patient months are reported as unanticipated ADEs.
Arm/Group | Early Recovery | Improvement | Non-improvement | Unassigned Based on Left Ventricular Ejection Fraction (LVEF)
All-Cause Mortality (participants affected / at risk) | 5/279 | 4/214 | 6/90 | 1/19
Serious Adverse Events (participants affected / at risk) | 0/279 | 1/214 | 0/90 | 0/19
Other Adverse Events (participants affected / at risk) | 8/279 | 14/214 | 3/90 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Recovery (N=279) | Improvement (N=214) | Non-improvement (N=90) | Unassigned Based on Left Ventricular Ejection Fraction (LVEF) (N=19)
Asystole with Inappropriate shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Inappropriate shock during asystole, occurring with hospitalization or death. Anticipated ADE.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Recovery (N=279) | Improvement (N=214) | Non-improvement (N=90) | Unassigned Based on Left Ventricular Ejection Fraction (LVEF) (N=19)
Skin irritation (Skin and subcutaneous tissue disorders) | 7 (8) | 12 (12) | 2 (2) | 0 (0) — Skin irritation with LifeVest
Discomfort (Product Issues) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Discomfort or pain from WCD
Inappropriate shock (Product Issues) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Inappropriate shock. Anticipated ADE
Frustration (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Frustration with alarms. Anticipated ADE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT03016754/Prot_SAP_000.pdf